CLINICAL TRIAL: NCT07262203
Title: Effectiveness of Diabetic Foot Exercises on Peripheral Vascular Status Among Patients With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Effect of Diabetic Foot Exercises on Peripheral Vascular Status in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Dr.Fahrun Nur Rosyid, S.Kep., Ns., M .Kes, Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMS-DFET2DM-2024
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Artery Disease (PAD); Diabetes Mellitus Type 2; Diabetic Foot Circulation Impairment
Keywords: diabetic foot exercises; peripheral vascular; ankle brachial index; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group controlled trial with two arms (intervention vs control). Participants were randomly allocated (1:1) using a card-shuffle randomization method. The intervention group performed a structured diabetic foot exercise program derived from Joslin Diabetes Center guidelines for three months (≈30 minutes/day, supervised monitoring), while the control group continued usual physical activity of comparable frequency and duration without the specific diabetic foot exercise program. Primary outcome (ankle-brachial index) measured at baseline and after 3 months using Doppler device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic Foot Exercise Intervention (Experimental): Participants performed a structured diabetic foot exercise program adapted from the Joslin Diabetes Center regimen. Exercises included quadriceps strengthening, balance exercises, ankle and foot mobility movements, and kicking exercises. The program was conducted for 3 months, approximately 30 minutes per day, with monitoring by the research team to maintain safety and adherence. All participants in this arm had type 2 diabetes mellitus. The primary outcome (ankle-brachial index) was measured at baseline and after 3 months.
  Interventions: Behavioral: Diabetic Foot Exercise Program
- Control - Usual Physical Activity (No Intervention): Participants continued their usual physical activities with similar recommended frequency and duration as the intervention group but did not receive the structured diabetic foot exercise program. They continued routine diabetes care and any prescribed DM medications. The control group served as a comparator to assess the effect of the diabetic foot exercise program on ankle-brachial index over 3 months

INTERVENTIONS:
Behavioral: Diabetic Foot Exercise Program — A structured diabetic foot exercise program adapted from the Joslin Diabetes Center protocol. The regimen includes quadriceps strengthening, balance exercises, ankle and foot mobility movements, and kicking exercises. Participants perform the exercises for approximately 30 minutes daily over 3 months under monitoring by the research team. The exercises aim to improve peripheral vascular status and lower-limb circulation. Ankle-brachial index is measured at baseline and after 3 months using a Doppler device
  Other Names: Diabetic Foot Exercises; Foot Exercise Regimen
  Arms: Diabetic Foot Exercise Intervention

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of diabetic foot exercises on peripheral vascular status among patients with type 2 diabetes mellitus. Peripheral artery disease is a common complication of diabetes and contributes to reduced mobility and increased risk of ulcers, ischemia, and amputation. Early identification and non-pharmacological interventions such as structured lower extremity exercises may help improve peripheral circulation.

In this study, 44 adults with type 2 diabetes mellitus who met the inclusion criteria were randomly assigned to either an intervention group receiving diabetic foot exercises or a control group performing regular physical activity of similar frequency and duration. The exercise protocol used in the intervention group was adapted from the Joslin Diabetes Center and included balance, strengthening, and ankle-foot mobility exercises. The intervention lasted for 3 months.

Peripheral vascular status was assessed using the ankle-brachial index (ABI) measured with a Doppler device at baseline and after 3 months. The study found that participants in the intervention group demonstrated a significant improvement in ABI values compared with the control group, indicating enhanced lower-limb blood flow.

This trial provides evidence that diabetic foot exercises are a simple, low-cost, and feasible intervention to improve peripheral vascular circulation in patients with type 2 diabetes mellitus, particularly in settings with limited resources.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted to determine the effectiveness of diabetic foot exercises in improving peripheral vascular status among patients with type 2 diabetes mellitus (T2DM). Diabetes mellitus is a chronic metabolic disorder associated with multiple vascular complications, including peripheral artery disease (PAD). PAD in diabetic patients is frequently asymptomatic during the early stages, yet it substantially increases the risk of ischemia, ulceration, and lower-limb amputation. Regular physical activity and targeted exercises have been shown to improve circulation and functional capacity. However, evidence regarding the effects of specific diabetic foot exercise programs on peripheral vascular status remains limited in Indonesia.

A total of 44 participants with T2DM were recruited from PERSADIA at Dr. Moewardi Hospital, Central Java, Indonesia. Participants were randomly assigned to either the treatment group (n = 22) or control group (n = 22) using a card-shuffle randomization method. Inclusion criteria included age above 50 years and a diagnosis of T2DM for at least 5 years. Exclusion criteria included inability to walk independently, lower extremity pain, severe arthritis, neurological or cardiovascular disorders, limited physical activity, or cognitive impairment. All participants provided written informed consent before enrollment.

The intervention consisted of a structured diabetic foot exercise program adapted from the Joslin Diabetes Center, involving quadriceps strengthening, balance exercises, ankle and foot mobility movements, and kicking exercises. Participants in the intervention group were instructed to perform the exercises daily for approximately 30 minutes over a period of 3 months, with monitoring to ensure safety. The control group participated in regular physical activity of similar duration and frequency but without the targeted diabetic foot exercise components.

Peripheral vascular status was assessed through the ankle-brachial index (ABI), using a Doppler device (ES-1000SPM, Hadeco, Japan). ABI measurements were taken at baseline and after 3 months of intervention, following standard procedures, including supine positioning and an initial rest period of five minutes. ABI categories followed established clinical thresholds: normal (0.90-1.30), mild impairment (0.70-0.89), moderate impairment (0.40-0.69), and severe impairment (<0.40).

Data analysis was performed using SPSS, employing paired t-tests for within-group comparisons and independent t-tests for between-group differences. The results demonstrated a significant improvement in ABI values in the intervention group (from 0.90 ± 0.05 to 0.96 ± 0.06), compared to minimal changes in the control group (from 0.90 ± 0.04 to 0.91 ± 0.05). These findings suggest that diabetic foot exercises can effectively enhance peripheral vascular function.

This study highlights that diabetic foot exercises offer a practical, low-cost, and accessible method for improving lower-extremity circulation in people with type 2 diabetes. Unlike intensive exercise programs requiring specialized equipment or supervision, this intervention is feasible for implementation in community settings and resource-limited environments. Although the study involved a relatively small sample size, the statistical power was acceptable, and the results align with previous evidence showing that lower extremity exercise improves vascular health.

Future studies with larger populations and longer follow-up periods are recommended to explore the long-term vascular and metabolic benefits of diabetic foot exercise programs

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged > 50 years
2. Diagnosed with Type 2 Diabetes Mellitus for ≥ 5 years
3. Able to walk independently
4. Willing to participate for the full 3-month intervention period
5. Provided written informed consent

Exclusion Criteria:

* patients who unable to walk independently, had lower limb pain, severe arthritis, cardiovascular or neurological disorders, limited physical activity, or cognitive dysfunction that impaired their ability to follow instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Ankle-Brachial Index (ABI) | Baseline and 3 months after intervention
  Ankle-Brachial Index (ABI) is measured using a handheld Doppler device (ES-1000SPM, Hadeco, Japan). ABI is calculated as the highest ankle systolic pressure (posterior tibial or dorsalis pedis) divided by the highest brachial systolic pressure. Measurements are taken in supine position after 5 minutes rest. ABI values reflect peripheral vascular status, categorized as normal (0.90-1.30), mild (0.70-0.89), moderate (0.40-0.69), and severe (<0.40). Primary analysis compares the change in ABI from baseline to 3 months between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Faculty of Health Sciences FIK UMS, Principal Investigator — Universitas Muhammadiyah Surakarta
Locations (1):
- RSUD Dr. Moewardi Surakarta, Surakarta, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The researchers do not plan to share individual participant data because the dataset contains sensitive health information and no data-sharing repository has been prepared for this study.